CLINICAL TRIAL: NCT02765919
Title: Study of Two Fractions Versus Three Fractions High Dose Rate Brachytherapy in Locally Advanced Carcinoma of Uterine Cervix After Pelvic Concurrent Chemoradiotherapy - a Randomized Controlled Trial
Brief Title: A Randomised Controlled Trial Between Two Different HDR Brachytherapy Schedule in Locally Advanced Carcinoma of Uterine Cervix
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr. Israt Jahan, Resident,Dept. of Oncology,BSMMU, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1356
Record Dates: First submitted 2016-05-05; First posted 2016-05-09 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Squamous Cell Carcinoma of Cervix
Keywords: Carcinoma cervix; RCT(randomised controlled trial); 9 Gray; Brachytherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiation HDR Brachytherapy 9 Gy (Experimental): High dose rate (HDR) Brachytherapy of weekly 9 Gray in two fractions in two weeks after 50 Gray of EBRT in 2 Gray per fraction of 5 weeks with chemotherapy cisplatin 40 mg /m2 weekly for five weeks in locally advanced carcinoma cervix
  Interventions: Radiation: HDR Brachytherapy of 9 Gy in 2 fractions
- Radiation HDR Brachytherapy 7 Gy (Active Comparator): High dose rate (HDR) brachytherapy of weekly 7 Gray in three fractions in three weeks after 50 Gray EBRT of 2 Gray per fraction of 25 fractions concurrently with weekly chemotherapy cisplatin40 mg /m2 in five weeks in locally advanced carcinoma cervix
  Interventions: Radiation: HDR Brachytherapy of 7 Gy in 3 fractions

INTERVENTIONS:
Radiation: HDR Brachytherapy of 9 Gy in 2 fractions — Two fractions of HDR brachytherapy following standard dose CCRT in locally advanced carcinoma cervix
  Arms: Radiation HDR Brachytherapy 9 Gy
Radiation: HDR Brachytherapy of 7 Gy in 3 fractions — Three fractions of HDR Brachytherapy following standard dose CCRT in locally advanced carcinoma cervix
  Arms: Radiation HDR Brachytherapy 7 Gy

SUMMARY:
The purpose of this study is to compare two different brachytherapy treatment option in locally advanced carcinoma of uterine cervix. Brachytherapy of two fractions of 9 Gy is effective in locoregional control and more convenient in terms of cost and time than 7 Gy brachytherapy of 3 fractions in management of locally advanced carcinoma of cervix.

DETAILED DESCRIPTION:
Cervical cancer is the second most common cancer among women worldwide and is the commonest form of gynecolgic malignancy in Bangladesh.Radiotherapy in the form of external beam radiotherapy combined with intracavitary Brachytherapy is the accepted definitive mode of treatment.Limiting the number of high dose rate(HDR) Brachytherapy has the potential benefit of improving patient compliance and reducing treatment cost and duration.The aim of this study is to compare the treatment outcome and acute complications following treatment with 9 Gray (Gy) in two fractions of brachytherapy with standard EBRT in locally advanced carcinoma of cervix.

EBRT will be delivered by a cobalt 60 teletherapy unit to a prescribed dose of 50 Gy in 25 fractions of 2 Gy per fraction and 5 days a week over a period of 5 weeks concurrent with inj. Cisplatin 40 mg/meter square weekly for 5 weeks.The patients will be then randomised into two arms of HDR brachytherapy,either 9Gy in 2 fractions or 7 Gy in 3 fractions.All patients will be followed up as per guideline for 6 months.The treatment related toxicity will be measured by Common Toxicity Criteria(Common terminology criteria for adverse events v.3.0).

All the relevant collected data will be compiled on a master chart and then statistical analysis of the results will be obtained by using SPSS 17.The data will be analysed using Chi square test and T test.Significant value will be decided at a level of 0.05 in two tailed tests.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced carcinoma cervix (stage 2b - 4a)
* Histopathology squamous cell carcinoma

Exclusion Criteria:

* Previous history of malignancy
* Previously treated with radiotherapy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-07; Primary Completion 2016-12 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Reduction of tumor size in cervix | Six month
  Comparison of pre treatment tumor size with post treatment tumor

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Abdul Bari, MBBS,MPhil, Study Director — Associate Professor,dept.of Oncology,BSMMU
Locations (1):
- BSM Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Patel FD, Rai B, Mallick I, Sharma SC. High-dose-rate brachytherapy in uterine cervical carcinoma. Int J Radiat Oncol Biol Phys. 2005 May 1;62(1):125-30. doi: 10.1016/j.ijrobp.2004.09.017. PMID 15850912
- See also: Related Info — http://www.bsmmu.edu.bd